CLINICAL TRIAL: NCT06937788
Title: Pragmatic Replication of the Heads Up Head-to-head Study of Upadacitinib and Dupilumab With TREATgermany Registry Data
Brief Title: Replication of the Heads Up Atopic Dermatitis Trial With Registry Data
Acronym: Re-HU-TREAT
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: TTE_101_TREATGer
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
Keywords: observational; target trial emulation; dupilumab; upadacitinib
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib; dupilumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- Upadacitinib (treatment group)
  Interventions: Drug: Upadacitinib
- Dupilumab (active comparator)
  Interventions: Biological: Dupilumab

INTERVENTIONS:
Drug: Upadacitinib — 30 mg tablet daily
  Groups: Upadacitinib (treatment group)
Biological: Dupilumab — 300 mg injection every other week
  Groups: Dupilumab (active comparator)

SUMMARY:
The goal is the replication of the primary outcome (EASI 75 at week 16) of the Heads Up trial (Blauvelt, A, Teixeira, H, Simpson, E et al (2021) doi:10.1001/jamadermatol.2021.3023) and the evaluation of the patient reported outcomes (POEM, DLQI and RECAP) in a head-to-head comparison of upadacitinib versus dupilumab treatment in moderate-to-severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is an inflammatory, multifactorial skin disease characterized by eczematous skin lesions, severe itching, and negative consequences on quality of life. The goal of this study is the replication of the primary outcome (Eczema Area and Severity Index (EASI) 75 at week 16) of the Heads Up trial and the evaluation of the patient reported outcomes (Patient-oriented Eczema Measure (POEM), Dermatologic Quality of Life Index (DLQI) and Recap of Atopic Eczema (RECAP)) that were not assessed in the Heads Up trial but are part of the recommendations by the Harmonising Outcome Measures for Eczema (HOME) initiative (Williams, HC, Schmitt, J, Thomas, KS et al (2022) doi:10.1016\j.jaci.2022.03.017) regarding core outcome sets in atopic dermatitis clinical trials. The core outcome set as defined by HOME encompasses the following domains (core outcome instruments): clinical signs (EASI), patient-reported symptoms (POEM and Peak Itch), long term control (RECAP) and quality of life (DLQI). The data basis is the TREATgermany registry (https://treatgermany.org/). TREATgermany is a national clinical registry for patients with moderate to severe AD. The physician and patient-reported outcomes are collected in about 60 clinics and private practices during routine care. Data of more than 2,400 patients is currently documented.

ELIGIBILITY:
Inclusion Criteria:

* Chronic AD with onset of symptoms at least 3 years prior to baseline
* Meets UK working party criteria
* EASI score ≥ 16
* ≥ 10% body surface area (BSA) of AD involvement at baseline ("therapy start") visit

Exclusion Criteria:

* contraindications according to upadacitinib or dupilumab labeling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with moderate to severe atopic dermatitis enrolled in the TREATgermany disease registry who are candidates for systemic therapy.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
POEM | baseline to month 6
  Mean POEM change

SECONDARY OUTCOMES:
DLQI | from baseline to month 6
  Mean DLQI change
RECAP | from baseline to month 6
  Mean RECAP change
EASI | from baseline to month 6
  Mean EASI change
NRS Itch (past 3 days) | from baseline to month 6
  Mean NRS Itch (past 3 days) change
NRS sleeping problems (past 3 days) | from baseline to month 6
  Mean NRS sleeping problems (past 3 days) change
EASI 75 | from baseline to month 6
  EASI 75 change

CONTACTS AND LOCATIONS:
Overall Officials: Jochen M Schmitt, Principal Investigator — Center for Evidence-based Healthcare, Medical Faculty and University Hospital Carl Gustav Carus, Technische Universität Dresden
Locations (1):
- Center for Evidence Based Health Care, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized data can be shared after receipt of data request outlining research question and data/variables needed and approval by TREATgermany prinicipal investigators.
Supporting Information: Study Protocol, ICF

REFERENCES:
- See also: TREATgermany website — https://treatgermany.org/